CLINICAL TRIAL: NCT07158138
Title: A Digitally Distributed Yoga Intervention in Prostate Cancer Rehabilitation (DigiYoga-P): Protocol for a Randomized Controlled Trial
Brief Title: A Digitally Distributed Yoga Intervention in Prostate Cancer Rehabilitation : Protocol for a Randomized Controlled Trial
Acronym: Digiyoga-P
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Dnr 2025-02611-01
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer Patients
Keywords: RCT; rehabilitation; yoga; Digital; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled multicenter study, where participants are randomized to an internet-based yoga intervention or a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Recieves a digital yoga intervention
  Interventions: Other: Digital yoga intervention
- Controllgroup (No Intervention): Recieves usual care

INTERVENTIONS:
Other: Digital yoga intervention — Digital yoga intervention
  Arms: Intervention group

SUMMARY:
Prostate cancer and its treatment can affect psychological, physical, and social quality of life. The most common side effects of the disease and treatment are bowel and urinary problems, sexual issues, and reduced quality of life. These issues can be alleviated with proper treatment and rehabilitation. Stress has been shown to be a significant factor in reduced quality of life.

The overall aim of the research project is to evaluate and compare the effect of an internet-based yoga intervention for individuals diagnosed with prostate cancer with a control group receiving standard care regarding stress, urinary incontinence, blood pressure, and quality of life. Additional objectives include describing cost-effectiveness and the experience of participating in an internet-based yoga intervention at home.

Scientific Questions Does internet-based yoga have any effect on stress, urinary incontinence, blood pressure, and quality of life compared to standard care? Is internet-based yoga a cost-effective intervention from the perspective of healthcare and society compared to standard care? How feasible is internet-based yoga, and how do participants perceive it? Does blood pressure change due to digital yoga, and does the effect persist after one year? Do participants in the intervention group continue practicing yoga after the intervention ends?

DETAILED DESCRIPTION:
There are no studies evaluating the effect of digital yoga in individuals diagnosed with prostate cancer.

The study is a randomized controlled multicenter study, where participants are randomized to an internet-based yoga intervention or a control group.

Study Participants Inclusion criteria are men diagnosed with prostate cancer without signs of metastatic disease, treated with curative intent.

Recruitment Participants are recruited through urology clinics and patient associations nationwide, as well as through social media such as Facebook and Instagram, and physical platforms such as bulletin boards and conferences. . receives standard care: standardized information about the importance of physical activity is included in the patients' care plan, which is offered to all prostate cancer patients. A Pilot Study A pilot study with five participants will be conducted before the intervention starts. The purpose of the pilot study is to test the yoga program. The pilot study will be evaluated through focus groups and individual interviews.

Data Collection Data is collected at baseline, within two months of diagnosis, after 3 and 6 months, and after 1 (and 2) years. An overview of the data collection schedule is shown in Appendix 2a.

Instruments for Patient-Reported Outcome Measures

* The Perceived Stress Scale measures general stress and coping capacity. The instrument is validated in a Swedish population and has 14 questions. Response options are: almost never, sometimes, fairly often, or very often. The higher the score, the greater the reported stress.
* EORTC-QLQ30 and the prostate cancer module measure health-related quality of life (HRQoL), consisting of 30 questions grouped into six scales: global health status, physical function, role function, emotional function, cognitive function, and social function. The prostate cancer module consists of 25 additional prostate cancer-specific questions.
* EuroQol-5D is a generic standardized instrument for measuring health-related quality of life, which is the basis for the health economic calculation. It includes 5 questions. The The Expanded Prostate Cancer Index Composite questionnaire with 26 questions developed to measure the quality of life in patients with prostate cancer and previously used in Sweden .

Additional Data Collection Basic data: Age, gender, marital status, occupation, sick leave, phone number, email address, postal address, yoga experience.

Disease-related data: Diagnosis date, planned treatment, previous illnesses (comorbidity according to Charlson comorbidity index). Other: Changes in treatment and additional leaves

Blood Pressure Measurement Home blood pressure measurement will be done wit.h the OMROM blood pressure monitor (Blood pressure monitor from Omron - Best in test Omron (omron-sverige.se)) sent to study participants and kept if the person completes the data collection. Home blood pressure measurement is a reliable method used in Region Örebro County and eliminates the suspicion of white coat effect, i.e., stress during medical visits. Research participants are expected to check their blood pressure morning and evening every day for a week at 4 occasions: inclusion week, after 3, 6, and 12 months. An average value will then be calculated. At least 4 days of measurements will be accepted. Instructions for blood pressure measurement will be:

* Sit and rest for 5 minutes
* Measure blood pressure sitting with the arm resting on a table.
* Measure morning and evening, two measurements with 1-2 minutes interval
* Register blood pressure through the email you received

Yoga Activity All study participants (both control and intervention) register how much yoga they have practiced each week through a digital survey. Medical and other clinical data: will be collected from medical records and from the Information Network for Cancer (INCA) regarding treatment, dose intensity, toxicity, and side effects according to NCI-CTC 4.0, as well as time to relapse and survival.

Data Storage Electronic data storage: All collected data is handled according to Region Örebro County's routines for research data and the information management plan for research documents. Collected data is stored pseudonymized on a dedicated storage area for research data, FoU Drive, which is adapted to requirements for handling research data containing sensitive personal information. FoU Drive is located in Region Örebro County's own data center and is part of a central file server solution with redundancy, backup, and logging according to the region's routines. Data collection for surveys is done electronically through SmartTrial, an electronic support system for collecting research data in clinical studies. The database is provided by Region Örebro County and the security in the system is compliant with regulations for storing sensitive data. Regular backups are made to secure data. Logging into all levels of the system requires two passwords. Participants need a login to register their responses. SmartTrial sends text messages and emails to remind participants to log in and complete surveys. Participants who prefer paper surveys will receive them by mail along with a prepaid return envelope. Paper data will be stored at the research center where only the research team has access to the data.

Health Economic Assessment Health economic assessment will be conducted from both a healthcare perspective and a societal perspective. Cost-effectiveness will be presented as the incremental cost per quality-adjusted life year (QALY), but also as a probability of cost-effectiveness compared to standard care. The main components of the analysis are additional costs or savings of interventions and changes in QALY. Savings can be reduced sick leave (less production losses) or healthcare consumption. QALY will be estimated using the EQ5D-5L instrument, sick leave time collected through questionnaires to participants, and healthcare consumption will be retrieved from patient records.

Experience of Internet-Based Yoga The experience of participating in the internet-based yoga intervention will be described through a study with qualitative methods where 15-20 patients are interviewed about their experience of participating in a web-based yoga intervention. Interview questions: Main question: How has it been to participate in a yoga class online? Complementary questions: What have you experienced as positive? What have you experienced as negative? How have you experienced the group practicing yoga simultaneously? How has your stress level been affected by yoga? The interviews will be transcribed verbatim and then analyzed with qualitative content analysis.

Intervention Fidelity Adherence to the project's method is regularly monitored during the study. The intervention responsible researcher has regular contact with the instructors and ensures that the program is followed. The methodology for data collection has been tested in the previous study Digiyogacare, which included women operated for breast cancer 26.

All yoga instructors have more than 300 hours of experience as yoga instructors and undergo training that includes study design, diagnosis, yoga program with possible adaptations.

Monitoring Side Effects and Dropouts Patients are informed to report any side effects and, if possible, the reasons for not completing the study will be recorded and later presented.

Significance for the Research Field Previous research has shown that live yoga for prostate cancer has a positive effect on fatigue, urinary and sexual function, and improved quality of life. There are few studies in the area, and it is unclear if the same effects can be achieved with digital yoga. Digiyoga-P is a randomized controlled study designed to determine if digital yoga is effective rehabilitation for the patient group. The methodology with digital yoga has previously been tested and refined by parts of the research team through a study of another diagnosis group, women operated for breast cancer in the research project Digiyogacare: Digitally distributed Yoga Intervention in Breast Cancer Rehabilitation 26. The preliminary analysis shows good results, and the project's infrastructure is well established and can largely be used in a prostate cancer context. Now the yoga intervention is adapted to the prostate cancer-related issues, including pelvic floor strengthening movements. The knowledge gap that the project fills is: What effect does digital yoga have for men diagnosed and treated with prostate cancer? Does it affect stress, urinary incontinence, blood pressure, and quality of life, and is any effect lasting? Is internet-based yoga cost-effective? How feasible is it, and how do participants perceive internet-based yoga? Do the intervention group continue practicing yoga even after the intervention ends?

Patient Benefit Common issues associated with prostate cancer are stress, bowel and urinary problems, sexual issues, and reduced quality of life. These problems can be alleviated with proper rehabilitation. Having to travel to the hospital for rehabilitation reduces accessibility for patients living far from the hospital. It can also be overwhelming to travel for treatments and rehabilitation. This study investigates whether internet-based yoga is a feasible form of rehabilitation that can contribute to equal rehabilitation regardless of the place of residence. Yoga for men has become increasingly relevant and media-covered in recent years, and therefore we believe it will be an attractive rehabilitation for men treated for prostate cancer. If side effects of diagnosis and treatment can be alleviated for the large group of prostate cancer patients, well-being can increase, and the pressure on healthcare can be reduced.

ELIGIBILITY:
Inclusion Criteria: are men diagnosed with prostate cancer without signs of metastatic disease, treated with curative intent. They should be Swedish-speaking and literate. Participants can be included within two months of diagnosis

-

Exclusion Criteria:

* are individuals under active surveillance or with advanced disease.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-01-10 (Estimated); Study Completion 2030-01-10 (Estimated)

PRIMARY OUTCOMES:
Does internet-based yoga have any effect on stress compared to standard care? | From enrollment to 12 months
  • The Perceived Stress Scale (PSS)20 measures general stress and coping capacity. The instrument is validated in a Swedish population and has 14 questions. Response options are: almost never, sometimes, fairly often, or very often. The higher the score, the greater the reported stress.
Stress | From enrollment to 12 months
  The Perceived Stress Scale (PSS)20 measures general stress and coping capacity. The instrument is validated in a Swedish population and has 14 questions. Response options are: almost never, sometimes, fairly often, or very often. The higher the score, the greater the reported stress.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Ohlsson-Nevo, Principal Investigator — USÖ
Locations (1):
- University Health Care Center, Örebro, Region Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No